CLINICAL TRIAL: NCT02669459
Title: A Randomized, Single Blinded Trial to Evaluate the Efficacy of Imiquimod in Women With Residual/Recurrent Cervical Intraepithelial Neoplasia (CIN) After Previous Treatment
Brief Title: Imiquimod Treatment of Residual or Recurrent CIN Lesions: a Study Protocol
Acronym: TopIC-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Maastricht University Medical Center (Other); Meander Medisch Centrum (Other); Albert Schweitzer Hospital (Other); Sint Franciscus Gasthuis (Other); Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, A.J.M. van de Sande, A. van de Sande, MD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL 53792.078.15; 2015-002308-10 (EudraCT Number)
Record Dates: First submitted 2016-01-15; First posted 2016-02-01 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Cervical Intraepithelial Neoplasia; Imiquimod; Human papillomavirus; quality of life; biological markers
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LLETZ (Active Comparator): LLETZ (Large Loop excision of the transformation zone) treatment conform current guidelines, which is also the current gold standard in the Netherlands
  Interventions: Procedure: LLETZ
- Imiquimod 5% cream (Other): intervention group
  Interventions: Drug: Imiquimod

INTERVENTIONS:
Drug: Imiquimod — 12,5 mg imiquimod three times per week during 16 weeks
  Other Names: aldara
  Arms: Imiquimod 5% cream
Procedure: LLETZ — surgical treatment for CIN, current gold standard
  Other Names: Large Loop Excision of the transformation zone
  Arms: LLETZ

SUMMARY:
The purpose of this study is to investigate if imiquimod can be used as a non-invasive option in the treatment of residual/recurrent CIN lesions.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE CIN Cervical dysplasia is caused by HPV and most common in women of reproductive age. Cervical dysplasia is known to be a precancerous stage of cervical cancer, where cervical cancer is the fourth most common cancer worldwide in women. Treatment of moderate to severe dysplasia is often still surgical and aimed at eliminating the affected part of the transformation zone. There are different type of surgical treatments (Large Loop excision of the transformation zone (LLETZ), knife cone biopsy, laser conisation), which have around 90% success rate. Historically moderate and severe dysplasia were treated with cold knife biopsy. Nevertheless, with deep cones hemorrhage, infection and postprocedure stenosis were reported. LLETZ seems to be a good alternative. It can be performed under local anesthesia, is cheaper, less painful and seem to have less short and long term morbidity. In outcome LETTZ has a similar risk in residual disease compared to cold knife cone. LLETZ is therefore the golden standard for treating cervical dysplasia nowadays. Still, there is uncertainty about the effects of LLETZ on short and long term in terms of recurrence, fertility and future pregnancy outcomes. Women diagnosed with CIN are usually at their reproductive age, so effects on future fertility and pregnancy are a concern. Women with a shorter time interval from LLETZ to pregnancy seem to have an increased risk for spontaneous abortion[6]. Also there is contradicting evidence on the presumed higher risk on preterm delivery and low birth weight. One study reported a 10 fold higher risk for preterm deliveries after more than one conisation procedure in women with cervical dysplasia. Furthermore, a recent study showed a higher subfertility rate with patients who underwent cervical surgery. Systematic review and meta-analysis reported on LLETZ for CIN also showed an increased rate of preterm delivery (<32wks RR 1.98, 95% CI 1.31-2.98; <28wks RR 2.33, 95% CI 1.84-2.94), premature rupture of the membranes (RR 1.88, 95% CI 1.54-2.29) and low birth weight (<2,500g RR 2.48, 95% CI 1.75-3.51) Apart from reproductive arguments there is an ongoing debate about the longterm outcome after treatment with surgical excision. Several studies show a recurrence rate of CIN 2-3 after treatment of 15-22 % within 2 years. Margin involvement seemed to be a risk factor for developing residual or recurrent cervical dysplasia Moreover, even after adequate treatment and follow up with normal smear results, patients who were treated for cervical intraepithelial dysplasia seem to have an excessive risk of cervical cancer compared to patients with normal primary smear test results. This risk is even almost 25 times higher in patients with abnormal smear test results than in patients with normal smear test results after treatment. Recent studies found that most women with residual or recurrent disease test positive for HPV after treatment. Possibly this could be a tool for risk stratification in the follow up after treatment. Also, this could raise the question if there is a need to treat HPV instead of treating the consequences of HPV (removing the transformation zone). Especially in patients with recurrent or residual disease.

Evidence for the involvement of Human Papilloma Virus in CIN Human Papilloma Virus (HPV) is the cause of pre-cancerous abnormalities of the cervix. HPV has over 100 subtypes and is present in over 95% of pre-invasive and invasive squamous carcinomas of the cervix. Some researchers state that HPV negative cervical cancer does not exist. Certain serotypes are associated with a high risk for progression to malignancy and more often found in cervical cancer. This are HPV type 16, 18, 31, 33, 35, 45, 52, and 58.

There is evidence that earlier detection of high stage CIN lesions (CIN 3) will be accomplished by screening with HPV DNA tests other than cytology alone.

Rationale Approximately 90% of the HPV is cleared after surgical treatment. Nonetheless, surgical treatment often deals more with the consequences instead of the cause of the disease. There is still a significant amount of women who will develop residual or recurrent disease. Recent publications show a higher risk of invasive cancer after treatment for cervical neoplasia grade 3 in comparison to the general population. Rebolj reported an incidence of 35,1 per 100000 years and 6,4 per 100000 years, respectively, led to an adjusted hazard ratio of 4,2 for periods after completed follow-up compared with periods after normal primary smear test results. Strander et al, showed an overall standardised incidence ratio for women with previous CIN grade 3 of 2,30 to develop invasive cervical carcinoma compared to the general population. Over time, there is a request for non-invasive treatment which treats HPV.

Young girls are vaccinated against HPV 16 and 18 nowadays. The current analysis show efficacy of almost 93% against CIN 2+associated with HPV-16/18 who had no evidence of oncogenic HPV infection on baseline. However only a 30% efficacy was seen against CIN2+ irrespective of HPV type in all women and 70% in the group who had no evidence of oncogenic HPV infection on baseline. For CIN3+ these numbers are 33% in the whole group and 87% in the HPV negative group. Vaccine efficacy against CIN2+ associated with 12 nonvaccine oncogenic types was 54%. Another problem is the vaccination uptake along young women. Since the reality is still that many women could or would not get vaccinated, primary prevention of HPV related diseases still has a long way to go.

STUDY DESIGN This is a randomized, single blinded, non-inferiority study in female patients with histologically recurrent/residual CIN of reproductive age after previous ablative treatment to evaluate the clinical and immunological effects of imiquimod. The estimated duration of the total study is 24 months, where a total of 433 patients will be included.

Patients will be randomized into one of two study groups:

1. Treatment with Imiquimod. Patients in this group will be treated with Imiquimod 5% for a total of 16 weeks.
2. LLETZ treatment (the standard treatment)

   STUDY POPULATION Population Inclusion of patients will take place in the Erasmus Medical Center Rotterdam, Meander hospital in Amersfoort, Albert Schweitzer Hospital in Dordrecht, Sint Franciscus hospital in Rotterdam, Catharina hospital in Eindhoven and Maastricht University Medical Centre and other hospitals in the Netherlands in the future. Patients will be drawn from colposcopy consultations. After qualifying for study participation based on pre-study procedures, patients will be randomized to receive either Imiquimod 5% cream or LLETZ (the standard treatment).

   Sample size calculation The regression rate of a second LLETZ procedure is estimated 63% in a retrospective cohort (data not published). The regression rate of CIN lesions after treatment with imiquimod was based upon the only study reporting on the regression rate after 16 weeks of imiquimod therapy of CIN. This study showed a regression rate of 73% in patients with primary CIN lesions. Since the effect could be lower in patients with residual or persistent CIN, we estimated the regression rate to be 60%. To calculate the required sample size in this two-proportions non-inferiority trial we assume that the probability of regression is 63% for the standard (LLETZ procedure) while it is 60% after treatment with imiquimod.

   Using a non-inferiority margin of 10% for the difference in proportions and a significance level (alpha) of 5%, a sample size of 174 per group is required to obtain a power of at least 80%. Allowing for 20% loss to follow-up the total required sample size is 433. [Chapter 4: Sample size calculations in clinical research (2nd edn). Shein-Chung Chow, Jun Shao and Hansheng Wang, Chapman & Hall/CRC, Boca Raton, FL, 2008 ] Because the uncertainty in the assumptions an interim analysis for futility will be performed by the DMC as soon as the primary outcome is available for 35 patients. This interim analysis is based on predictive power. That is the predicted probability of being able to prove non-inferiority given the results at the interim analysis. When the predictive power at this point is below 20% the trial will be stopped due to futility. Of course the DMC can always stop the trial due to safety concerns. The trial will never be stopped prematurely for efficacy so no alpha-adjustment is made.

   Description and justification of route of administration and dosage Imiquimod 5% cream will be administered in a vaginal applicator, containing 12,5 mg of Imiquimod (one sachet). The cream will be administrated three times per week before going to bed by the patients themselves. In case of uncomfortable reactions the application can be reduced twice or ones per week if side effects persist. When local side effects persist medication can be discontinued for one week.

   The following treatment protocol will be applied:

   - Treatment period for 16 weeks, in which 3 doses of 1 sachet (12,5 mg Imiquimod) will be applied three times per week.

   Preparation and labelling of Investigational Medicinal Product The organization of the preparation and labelling of imiquimod crème will be organized by the pharmacist of the Erasmus Medical Center. Preparation and labelling of the investigational medicinal products will be done according to the relevant GMP guidelines. The labels will be in Dutch for the Dutch centers. (according to the CCMO rules). Distribution and labelling of the study medication will be organized by the pharmacist of the Erasmus Medical Center.

   METHODS Randomisation, blinding and treatment allocation After signing the consent form, the patient will be randomized with the use of a computer program, in order to conceal the treatment allocation. Both doctor and patient will not know before randomization what treatment the patient will be allocated to. Study medication will be randomized according to a 1:1 ratio, such that there is 1 patient assigned to imiquimod for every patient on LLETZ. Randomisation will be performed in variable blocks. The study is single-blinded, which means only the pathologist will not be informed of the outcome randomization. Analysis will take place in intention-to-treat.

   Study procedures Week 0 for all patients

   The following procedures must be undertaken:
   * Informed consent signed
   * Assigning a study number
   * Confirmation of the in- and exclusion criteria
   * Collect demographic data
   * Relevant medical and surgical history
   * Quality of life questionnaire will be handed out
   * Urine pregnancy test if necessary. Contraception will be discussed and prescribed if necessary.
   * Dispense study medication and instruct the patient how to apply the imiquimod cream
   * Patients are randomized into one of two groups:

     -- Intervention group (12,5 mg imiquimod three times per week during 16 weeks)

     -- Standard treatment, consisting of LLETZ or CKC.
   * Make a new appointment for week 2 for the patients in the Imiquimod group
   * Make a new appointment for LLETZ treatment in the LLETZ group.

   Week 1, 2, 6,10, 11 and 12 for patients in the Imiquimod group

   After 1 week and 11 weeks there will be a telephone consultation. In this consultation the side effects, as experienced by patients, will be documented. After 2, 6, 10 and 12 weeks of treatment (+/-2 days) a study visit will be conducted. The following procedures must be undertaken:
   * Ascertain whether the patient has experienced any adverse events since the previous visit. This will be documented according to the Common Terminology Criteria for Adverse Events guidelines.
   * Ascertain whether the patient has used any concomitant medication or has any change in the concomitant medication
   * Collect and review the patient diary card to monitor compliance
   * At week 10 colposcopic examination (and biopsy if suspicion of invasive disease)
   * Dispense study medication
   * If necessary lower the imiquimod dose

   Week 0-1 In the LLETZ group: an appointment to perform the surgical procedure. After the procedure, follow up will be according to the dutch guidelines. This means cervical smears at 6, 12 and 24 months after the treatment with determination of HPV. If the patient has a PAP 2 or more or is carrying a high risk HPV during follow up, a colposcopy with biopsies will be performed to determine the CIN classification.

   Week 16 for patients in the Imiquimod group After 16 weeks of treatment (+/- 2 days) the fifth study visit will be conducted. The following procedures must be undertaken: - Ascertain whether the patient has experienced any adverse events since the previous visit by asking generally about patients health
   * Ascertain whether the patient has used any concomitant medication or has any change in the concomitant medication
   * Collect and review the patient diary card to monitor compliance
   * Collect study medication
   * Make a new appointment for week 26.

   Week 26 After 26 weeks (+/- days) the sixth study visit for the imiquimod group and will be conducted.

   The following procedures must be undertaken:

   In the Imiquimod group

   - Ascertain whether the patient has experienced any adverse events since the previous visit according to the Common Terminology Criteria for Adverse Events guidelines.

   - Ascertain whether the patient has used any concomitant medication or has any change in the concomitant medication

   - Colposcopic examination and biopsy for histology in the Imiquimod group

   - Surgical treatment will be performed in case of progression or stabilization of disease.

   There will be a conservative treatment with follow up of cervical smears in cases of regression of disease.

   - Quality of life questionnaire will be handed out.

   - Cervix cytology and HPV typing.
   * Make a new appointment for month 6 of follow-up

   Month 6 after treatment

   After 6 months the following procedures must be undertaken:

   - Quality of life questionnaire
   * Cervix smears and HPV determination

   Month 12 after treatment

   After 12 months the following procedures must be undertaken:
   * Quality of life questionnaire
   * Cervix smears and HPV determination

   Month 24 after treatment After 12 months the final study visit will be conducted. The following procedures must be undertaken: - Cervical smears and HPV determination - Informed consent for retrieving information about outcome of cervical cytology or HPV testing from national prevention approximately 5 years after treatment. This information will be retrieved from the national databank, general practitioner or patient itself.

   A biopsy of the cervix has been taken within 3 months prior of the start of the trial, together with a frozen tissue for HPV typing. Patients with a histologically proven CIN 2 and CIN 3 or persistent CIN 1 after previous treatment will be informed of the study and given written information about it. When assessed for eligibility the patient will be asked to give written informed consent to inclusion in the trial.

   Every visit, a questionnaire will be filled in to evaluate symptoms and adverse events. Side effects and adverse events will be documented according to Common Terminology Criteria for Adverse Events guidelines during the checkups. Patients are also instructed to report adverse events immediately and visit the hospital if necessary. Diary card completion and dosing procedures will be reviewed at all treatment visits. Clinically significant abnormalities associated with adverse events will be followed. Because of unknown possible effects of imiquimod treatment, it is necessary to exclude pregnancy before enrolment in to the study. Moreover, contraception will be advised during the treatment period because of the unknown effects of Imiquimod during pregnancy. Many CIN-patients are also diagnosed with VIN and VAIN lesions, so at colposcopy also the vagina and vulva will be inspected and if necessary, taken biopsies. At 26 weeks (ten weeks after the treatment period) a biopsy will be taken of the area of the cervical lesion judged most abnormal and a HPV DNA assay will be conducted. Also cytology will be taken. If the classification of CIN is increased or stabilised, LLETZ will be performed. Patients with PAP 3B or more at cytology and colposcopic suspicion of CIN1 or less will also be treated with LLETZ to rule out invasive disease of another location than the biopsy taken. Patients with regression of the CIN classification of the lesion (with cytology PAP3A or less) will be treated conservative and will be followed up in the same schedule as patients after LLETZ.

   At 6 and 18 months after finishing treatment cytology will be taken as follow-up. When there is cytology is abnormal a colposcopy will be performed. When recurrence of CIN 2 or 3 or invasive disease is suspected at another biopsy will be taken. Further treatment will be according to the expertise of the treating physician.

   To evaluate the quality of life the following questionnaires will be used.

<!-- -->

1. Medical Outcomes Study 36-Item Short-Form General Health Survey (RAND 36), to access generic health-related quality of life.
2. European Organization for Research and Treatment of Cancer (EORTC) quality-of-life questionnaire: QLQ-C30, to assess cancer-specific health-related quality of life.
3. European Organization for Research and Treatment of Cancer (EORTC) quality-of-life questionnaire: QLQ-CX24, to assess cervical specific quality of life, including sexual functioning.

   Patient withdrawal or discontinuation

   Following treatment initiation, each patient's trial participation will end when one of the following occurs:
   * Patient has completed all study procedures including 16 weeks of treatment, and follow-up visit at 26 weeks, 12 and 24 months.
   * Patient discontinues study participation prior to completion of all study procedures.

   Patients may withdraw themselves from the study at any time, or be withdrawn by the investigator, without prejudice to their future medical care. The investigator can decide to withdraw a subject from the study for urgent medical reasons.

   Specific criteria for withdrawal Patients who become pregnant during the study will be immediately discontinued from further study participation and will complete all withdrawal procedure prior to discontinuation. The investigator will record the reason for withdrawal and the date of such occurrence on the patient status record.

   Replacement of individual subjects after withdrawal Withdrawn individuals will not be replaced.

   Follow-up of subjects withdrawn from treatment If a patient discontinues the study due to an adverse event or laboratory abnormality, the investigator will follow the patient until the adverse event has resolved or reached a stable condition. In any case of withdrawal the patients will be offered the treatment of recurrent/residual CIN which will be advised by the treating physician of the patient. They will be followed up by the current guidelines.

   Premature termination of the study If any unexpected severe side effects occur, the study will be prematurely terminated after advise of the DMSB. The METC will be informed.

   SAFETY REPORTING Section 10 WMO event In accordance to section 10, subsection 1, of the WMO, the investigator will inform the subjects and the reviewing accredited METC if anything occurs, on the basis of which it appears that the disadvantages of participation may be significantly greater than was foreseen in the research proposal. The study will then be suspended pending further review by the accredited Ethical Board, except insofar as suspension would jeopardise the subjects' health. The investigator will take care that all subjects are kept informed.

   Adverse and serious adverse events Adverse events (AEs) are defined as any undesirable experience occurring to a subject during a clinical trial, whether or not considered related to the investigational drug. All adverse events reported spontaneously by the subject or observed by the investigator or his staff will be recorded. A Serious Adverse Event (SAE) is any untoward medical occurrence or effect that at any dose

   - results in death;

   - is life threatening (at the time of the event);

   - requires hospitalisation or prolongation of existing inpatients' hospitalisation;

   - results in persistent or significant disability or incapacity;

   - is a congenital anomaly or birth defect;

   - is a new event of the trial likely to affect the safety of the subjects, such as an unexpected outcome of an adverse reaction, lack of efficacy of an IMP used for the treatment of a life threatening disease, major safety finding from a newly completed animal study, etc. All SAEs will be reported to the accredited METC that approved the protocol, according to the requirements of that METC.

   Suspected unexpected serious adverse reactions (SUSAR) Adverse reactions are all untoward and unintended responses to an investigational product related to any dose administered.

   Unexpected adverse reactions are SUSARs if the following three conditions are met:

1. the event must be serious. 2. There must be a certain degree of probability that the event is harmful and an undesirable reaction to the medicinal product under investigation, regardless of the administered dose.

3. The adverse reaction must be unexpected, that is to say, the nature and the severity of the adverse reaction are not in agreement with the product information as recorded in:

-- Summary of Product Characteristics (SPC) for an authorised medicinal product;

-- Investigator's Brochure for an unauthorised medicinal product.

The sponsor will report expedited the following SUSARs to the METC:

* SUSARs that have arisen in the clinical trial that was assessed by the METC;
* SUSARs that have arisen in other clinical trial of the same sponsor and with the same medicinal product, and that could have consequences for the safety of the subjects involved in the clinical trial that was assessed by the METC. The remaining SUSARs are recorded in an overview list (line-listing) that will be submitted once every half year to the METC. This line-listing provides an overview of all SUSARs from the study medicine, accompanied by a brief report highlighting the main points of concern.

The sponsor will report expedited all SUSARs to the competent authority, the Medicine Evaluation Board and the competent authorities in other Member States. The expedited reporting will occur not later than 15 days after the sponsor has first knowledge of the adverse reactions. For fatal or life threatening cases the term will be maximal 7 days for a preliminary report with another 8 days for completion of the report.

Annual safety report

In addition to the expedited reporting of SUSARs, the sponsor will submit, once a year throughout the clinical trial, a safety report to the accredited METC, competent authority, Medicine Evaluation Board and competent authorities of the concerned Member States. This safety report consists of:

* a list of all suspected (unexpected or expected) serious adverse reactions, along with an aggregated summary table of all reported serious adverse reactions, ordered by organ system, per study;
* a report concerning the safety of the subjects, consisting of a complete safety analysis and an evaluation of the balance between the efficacy and the harmfulness of the medicine under investigation.

Follow-up of adverse events All adverse events will be followed until they have abated, or until a stable situation has been reached. Depending on the event, follow up may require additional tests or medical procedures as indicated, and/or referral to the general physician or a medical specialist.

STATISTICAL ANALYSIS Statistical analysis is performed with SPSS (SPSS Inc., Chicago, IL) for the individual features studies.

Primary study parameter Analysis will be done according to the non-inferiority principle to show that imiquimod is not worse than an existing treatment (LLETZ). To investigate efficacy we will perform a perprotocol analysis (although this is not the primary outcome of the study). The primary outcome is the difference between the probability of regression in the LLETZ and the imiquimod arms. The expected difference (LLETZ-imiquimod) will be calculated together with the 95% Aggresti confidence interval. If the upper bound of the interval lies below the noninferiority margin of 10% non-inferiority of the imiquimod treatment is assumed to be proved. Logistic analysis of potential confounders (age at diagnosis, CIN grade, number of previous treatments, smoking, HPV- subtype) will be performed. Withdrawn subjects will not be replaced. Analysis will be based on intention to treat protocol.

ETHICAL CONSIDERATIONS

Regulation statement This study will be conducted according to Good Clinical Practice (GCP), the Declaration of Helsinki (version 2004) and in accordance with the Medical Research Involving Human Subjects Act (WMO). The study will only be undertaken when fully approval of the protocol and patient information and consent form has been obtained from the appropriate Ethics Committee.

Recruitment and consent Recruitment Inclusion of patients will take place at the Erasmus Medical Center in Rotterdam, Meander Hospital in Amersfoort and Albert Schweitzer Hospital in Dordrecht. More hospitals can participate if they perform colposcopy and LLETZ in their center. Patients will be informed of the study after diagnosed with cervical dysplasia grade 2-3 proved by biopsy. They will receive the patient information and an informed consent form. On the outpatient clinic patients will be granted time to ask questions about the procedures. During this visit all procedures are explained and patients will be asked if they are willing to participate in the study. The patient will take written information home and will receive a next appointment to ask questions and to sign the inform consent.

Informed consent Prior to entering the study, the investigator will explain to each patient, the nature of the study, its purpose, procedures, expected duration, alternative therapy available, and the benefits and risks involved in study participation. Each patient will be informed of her right to withdraw from the study at any time without prejudice. After this explanation and before any study-specific procedures have been performed, the patient, as well as the investigator, will voluntarily sign and date an informed consent statement.

Benefits and risks assessment, group relatedness The possible benefit for the participating subject may be an effective treatment of their disease, which can lead to a complete clinical response of CIN and a total clearance of HPV. In contrast to surgical treatments (e.g. local excision) this treatment targets the cause of CIN, namely hrHPV. This may lead to a lower recurrence rate. Furthermore, the treatment is noninvasive and leaves the anatomy intact. Second, other HPV related disease like VAIN could be treated as well.

Risk and burden are linked to protocol procedures, such as biopsy sampling. Although these are routine procedures, carried out by medical qualified personnel, they may cause side effects or discomfort to the subject. However, it is expected that these procedures will generally be well tolerated.

In addition, since teratogenous effects of imiquimod are unknown, it is recommended that patients use adequate contraceptives during the study.

ADMINISTRATIVE ASPECTS AND PUBLICATION Handling and storage of data and documents Subject numbers will be assigned sequentially to subjects enrolled in the study. All data collected in this research protocol will be treated confidential and identified with the subject number not with the subjects name or address. A safety physician safeguards the investigational code All biopsies and serum samples will be stored in a secure location and will be kept for 15 years. All study records will also be archived in a safe and secure location. To verify the accuracy of the data, study records will be available to the representatives of the Dutch government (e.g. Inspection of Public Health) and members of the Ethical Board committee are allowed to inspect the quality of the accomplished research.

Monitoring and quality assurance The study was determined by the medical committee and through the medical plan of Erasmus medical center, as a study with a negligible risk. Determination of the risk analysis is enclosed. Monitoring will be done according to the current guidelines of the Erasmus Medical Center. For studies with a negligible risk, and annual visit will be performed by an external monitoring board.

Amendments Amendments are changes made to the research after a favourable opinion by the accredited METC has been given. All amendments will be notified to the METC that gave a favourable opinion.

A 'substantial amendment' is defined as an amendment to the terms of the METC application, or to the protocol or any other supporting documentation, that is likely to affect to a significant degree:

* the safety or physical or mental integrity of the subjects of the trial;
* the scientific value of the trial;
* the conduct or management of the trial; or
* the quality or safety of any intervention used in the trial.

All substantial amendments will be notified to the METC and to the competent authority.

Non-substantial amendments will not be notified to the accredited METC and the competent authority, but will be recorded and filed by the sponsor.

Annual progress report The investigator will submit a summary of the progress of the trial to the accredited METC once a year. Information will be provided on the date of inclusion of the first subject, numbers of subjects included and numbers of subjects that have completed the trial, serious adverse events/ serious adverse reactions, other problems, and amendments.

End of study report The sponsor will notify the accredited METC and the competent authority of the end of the study within a period of 90 days. The end of the study is defined as the last patient's last visit (at 52 weeks).

In case the study is ended prematurely, the sponsor will notify the accredited METC and the competent authority within 15 days, including the reasons for the premature termination. Within one year after the end of the study, the investigator/sponsor will submit a final study report with the results of the study, including any publications/abstracts of the study, to the accredited METC and the Competent Authority.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CIN 2 or CIN 3, without invasion after previous surgical treatment at least 6 months before diagnosis.
* Histologically proven recurrent CIN 1 after previous surgical treatment at least 6 months before diagnosis. Persistent CIN 1 is defined as CIN 1 at least persistent for 6 months and proven with histology.
* The patient is willing to use a medically acceptable method of contraception throughout the study
* Women older than 18 years of age.

Exclusion Criteria:

* Pregnancy or lactation
* (Micro-)invasive carcinoma
* Past history of cervical cancer
* Hypersensitivity of any components of the formulation
* History of psoriasis or other inflammatory dermatosis of the vulva
* Immunodeficiency or treatment with immunosuppressive medication
* Insufficient understanding of the Dutch or English language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Reduction to normal cytology | 6 months after treatment

SECONDARY OUTCOMES:
Reduction to no dysplasia | 10 weeks after the treatment
  only Imiquimod group
presence or absence of HPV DNA in CIN lesions | presence in biopsy before start treatment, cervical smear 6 months after treatment
  Biopsy which is take prior to treatment for inclusion in the study
tolerability to the treatment/side effects | At 6 months, worst grade observed.
  Side effects (headache, fever, fatigue, myalgia, vaginal discharge, vaginal bleeding, vaginal pain/itch, vaginal swelling, other) noted in CTCAE grade (no side effects to grade 4)
tolerability to the treatment/side effects | At 6 months, worst grade observed.
  Side effects (headache, fever, fatigue, myalgia, vaginal discharge, vaginal bleeding, vaginal pain/itch, vaginal swelling, other) noted in VAS score (0-10)
quality of life | at inclusion for study, 6 and 12 months after start treatment
  QOL measured with RAND-36 scoring
quality of life | at inclusion for study, 6 and 12 months after start treatment
  QOL measured with QLQ-C30 scoring
quality of life | at inclusion for study, 6 and 12 months after start treatment
  QOL measured with QLQ-CX24 scoring
durability of the clinical response | PAP 1 at 12 and 24 months after the start treatment.
  Cervical smear taken at 12 and 24 months after start treatment in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Heleen van beekhuizen, MD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Result] Wright TC Jr, Gagnon S, Richart RM, Ferenczy A. Treatment of cervical intraepithelial neoplasia using the loop electrosurgical excision procedure. Obstet Gynecol. 1992 Feb;79(2):173-8. PMID 1731281
- [Result] Martin-Hirsch PL, Paraskevaidis E, Kitchener H. Surgery for cervical intraepithelial neoplasia. Cochrane Database Syst Rev. 2000;(2):CD001318. doi: 10.1002/14651858.CD001318. PMID 10796771
- [Result] Luesley DM, McCrum A, Terry PB, Wade-Evans T, Nicholson HO, Mylotte MJ, Emens JM, Jordan JA. Complications of cone biopsy related to the dimensions of the cone and the influence of prior colposcopic assessment. Br J Obstet Gynaecol. 1985 Feb;92(2):158-64. doi: 10.1111/j.1471-0528.1985.tb01068.x. PMID 3970895
- [Result] Sadek AL. Needle excision of the transformation zone: A new method for treatment of cervical intraepithelial neoplasia. Am J Obstet Gynecol. 2000 Apr;182(4):866-71. doi: 10.1016/s0002-9378(00)70337-1. PMID 10764464
- [Result] Conner SN, Cahill AG, Tuuli MG, Stamilio DM, Odibo AO, Roehl KA, Macones GA. Interval from loop electrosurgical excision procedure to pregnancy and pregnancy outcomes. Obstet Gynecol. 2013 Dec;122(6):1154-9. doi: 10.1097/01.AOG.0000435454.31850.79. PMID 24201682
- [Result] Jin G, LanLan Z, Li C, Dan Z. Pregnancy outcome following loop electrosurgical excision procedure (LEEP) a systematic review and meta-analysis. Arch Gynecol Obstet. 2014 Jan;289(1):85-99. doi: 10.1007/s00404-013-2955-0. Epub 2013 Jul 11. PMID 23843155
- [Result] Bevis KS, Biggio JR. Cervical conization and the risk of preterm delivery. Am J Obstet Gynecol. 2011 Jul;205(1):19-27. doi: 10.1016/j.ajog.2011.01.003. Epub 2011 Feb 23. PMID 21345402
- [Result] Ortoft G, Henriksen T, Hansen E, Petersen L. After conisation of the cervix, the perinatal mortality as a result of preterm delivery increases in subsequent pregnancy. BJOG. 2010 Feb;117(3):258-67. doi: 10.1111/j.1471-0528.2009.02438.x. Epub 2009 Nov 26. PMID 19943823
- [Result] Spracklen CN, Harland KK, Stegmann BJ, Saftlas AF. Cervical surgery for cervical intraepithelial neoplasia and prolonged time to conception of a live birth: a case-control study. BJOG. 2013 Jul;120(8):960-5. doi: 10.1111/1471-0528.12209. Epub 2013 Mar 14. PMID 23489374
- [Result] Serati M, Siesto G, Carollo S, Formenti G, Riva C, Cromi A, Ghezzi F. Risk factors for cervical intraepithelial neoplasia recurrence after conization: a 10-year study. Eur J Obstet Gynecol Reprod Biol. 2012 Nov;165(1):86-90. doi: 10.1016/j.ejogrb.2012.06.026. Epub 2012 Jul 6. PMID 22771223
- [Result] Rebolj M, Helmerhorst T, Habbema D, Looman C, Boer R, van Rosmalen J, van Ballegooijen M. Risk of cervical cancer after completed post-treatment follow-up of cervical intraepithelial neoplasia: population based cohort study. BMJ. 2012 Oct 31;345:e6855. doi: 10.1136/bmj.e6855. PMID 23117059
- [Result] Strander B, Andersson-Ellstrom A, Milsom I, Sparen P. Long term risk of invasive cancer after treatment for cervical intraepithelial neoplasia grade 3: population based cohort study. BMJ. 2007 Nov 24;335(7629):1077. doi: 10.1136/bmj.39363.471806.BE. Epub 2007 Oct 24. PMID 17959735
- [Result] McIndoe WA, McLean MR, Jones RW, Mullins PR. The invasive potential of carcinoma in situ of the cervix. Obstet Gynecol. 1984 Oct;64(4):451-8. PMID 6483293
- [Result] Ryu A, Nam K, Kwak J, Kim J, Jeon S. Early human papillomavirus testing predicts residual/recurrent disease after LEEP. J Gynecol Oncol. 2012 Oct;23(4):217-25. doi: 10.3802/jgo.2012.23.4.217. Epub 2012 Sep 19. PMID 23094124
- [Result] Cubie HA, Canham M, Moore C, Pedraza J, Graham C, Cuschieri K. Evaluation of commercial HPV assays in the context of post-treatment follow-up: Scottish Test of Cure Study (STOCS-H). J Clin Pathol. 2014 Jun;67(6):458-63. doi: 10.1136/jclinpath-2013-202014. Epub 2014 Jan 16. PMID 24436334
- [Result] Walboomers JM, Jacobs MV, Manos MM, Bosch FX, Kummer JA, Shah KV, Snijders PJ, Peto J, Meijer CJ, Munoz N. Human papillomavirus is a necessary cause of invasive cervical cancer worldwide. J Pathol. 1999 Sep;189(1):12-9. doi: 10.1002/(SICI)1096-9896(199909)189:13.0.CO;2-F. PMID 10451482
- [Result] de Sanjose S, Quint WG, Alemany L, Geraets DT, Klaustermeier JE, Lloveras B, Tous S, Felix A, Bravo LE, Shin HR, Vallejos CS, de Ruiz PA, Lima MA, Guimera N, Clavero O, Alejo M, Llombart-Bosch A, Cheng-Yang C, Tatti SA, Kasamatsu E, Iljazovic E, Odida M, Prado R, Seoud M, Grce M, Usubutun A, Jain A, Suarez GA, Lombardi LE, Banjo A, Menendez C, Domingo EJ, Velasco J, Nessa A, Chichareon SC, Qiao YL, Lerma E, Garland SM, Sasagawa T, Ferrera A, Hammouda D, Mariani L, Pelayo A, Steiner I, Oliva E, Meijer CJ, Al-Jassar WF, Cruz E, Wright TC, Puras A, Llave CL, Tzardi M, Agorastos T, Garcia-Barriola V, Clavel C, Ordi J, Andujar M, Castellsague X, Sanchez GI, Nowakowski AM, Bornstein J, Munoz N, Bosch FX; Retrospective International Survey and HPV Time Trends Study Group. Human papillomavirus genotype attribution in invasive cervical cancer: a retrospective cross-sectional worldwide study. Lancet Oncol. 2010 Nov;11(11):1048-56. doi: 10.1016/S1470-2045(10)70230-8. Epub 2010 Oct 15. PMID 20952254
- [Result] Bulkmans NW, Berkhof J, Rozendaal L, van Kemenade FJ, Boeke AJ, Bulk S, Voorhorst FJ, Verheijen RH, van Groningen K, Boon ME, Ruitinga W, van Ballegooijen M, Snijders PJ, Meijer CJ. Human papillomavirus DNA testing for the detection of cervical intraepithelial neoplasia grade 3 and cancer: 5-year follow-up of a randomised controlled implementation trial. Lancet. 2007 Nov 24;370(9601):1764-72. doi: 10.1016/S0140-6736(07)61450-0. Epub 2007 Oct 4. PMID 17919718
- [Result] Rijkaart DC, Berkhof J, Rozendaal L, van Kemenade FJ, Bulkmans NW, Heideman DA, Kenter GG, Cuzick J, Snijders PJ, Meijer CJ. Human papillomavirus testing for the detection of high-grade cervical intraepithelial neoplasia and cancer: final results of the POBASCAM randomised controlled trial. Lancet Oncol. 2012 Jan;13(1):78-88. doi: 10.1016/S1470-2045(11)70296-0. Epub 2011 Dec 14. PMID 22177579
- [Result] Moore EE, Danielewski JA, Garland SM, Tan J, Quinn MA, Stevens MP, Tabrizi SN. Clearance of human papillomavirus in women treated for cervical dysplasia. Obstet Gynecol. 2011 Jan;117(1):101-108. doi: 10.1097/AOG.0b013e3182020704. PMID 21173650
- [Result] Paavonen J, Naud P, Salmeron J, Wheeler CM, Chow SN, Apter D, Kitchener H, Castellsague X, Teixeira JC, Skinner SR, Hedrick J, Jaisamrarn U, Limson G, Garland S, Szarewski A, Romanowski B, Aoki FY, Schwarz TF, Poppe WA, Bosch FX, Jenkins D, Hardt K, Zahaf T, Descamps D, Struyf F, Lehtinen M, Dubin G; HPV PATRICIA Study Group. Efficacy of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine against cervical infection and precancer caused by oncogenic HPV types (PATRICIA): final analysis of a double-blind, randomised study in young women. Lancet. 2009 Jul 25;374(9686):301-14. doi: 10.1016/S0140-6736(09)61248-4. Epub 2009 Jul 6. PMID 19586656
- [Result] Grimm C, Polterauer S, Natter C, Rahhal J, Hefler L, Tempfer CB, Heinze G, Stary G, Reinthaller A, Speiser P. Treatment of cervical intraepithelial neoplasia with topical imiquimod: a randomized controlled trial. Obstet Gynecol. 2012 Jul;120(1):152-9. doi: 10.1097/AOG.0b013e31825bc6e8. PMID 22914404
- [Derived] van de Sande AJM, Koeneman MM, Gerestein CG, Kruse AJ, van Kemenade FJ, van Beekhuizen HJ. TOPical Imiquimod treatment of residual or recurrent cervical intraepithelial neoplasia (TOPIC-2 trial): a study protocol for a randomized controlled trial. BMC Cancer. 2018 Jun 15;18(1):655. doi: 10.1186/s12885-018-4510-7. PMID 29902979